CLINICAL TRIAL: NCT02845401
Title: "BeNEG-DO": A Study of Clinical Outcomes, Immunologic Correlates and Genetic Predictors After Treatment Withdrawal in e-Antigen Negative (HBeAg-) Chronic Hepatitis B Virus (HBV) Infection
Brief Title: The Hepatitis B e-Antigen Negative Disease - Directly Offered Study of Treatment Withdrawal in Patients With e-Antigen Negative Chronic HBV Infection (BeNEG-DO).
Acronym: BeNEG-DO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: California Pacific Medical Center Research Institute (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1R01DK103735-01A1 (NIH)
Record Dates: First submitted 2016-07-21; First posted 2016-07-27 (Estimated); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Chronic Hepatitis B Virus
Keywords: Viral; Hepatitis
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HBeAg-CHB patients who stop NA Therapy (Experimental): Patients with early antigen negative form of disease (HBeAg-CHB) who are already taking standard oral HBV antiviral therapy for at least 192 weeks that stop treatment.
  Intervention: Cases will stop antiviral therapy
  Interventions: Other: Stop NA therapy
- HBeAg-CHB patients continue NA Therapy (No Intervention): Patients with early antigen negative form of disease (HBeAg-CHB) who are already taking standard oral HBV antiviral therapy for at least 192 weeks that continue to stay on treatment.
  Intervention: None. Controls will continue antiviral therapy.

INTERVENTIONS:
Other: Stop NA therapy — Cases will stop antiviral therapy
  Arms: HBeAg-CHB patients who stop NA Therapy

SUMMARY:
The investigators' research is aimed at developing more effective, finite approaches for managing individual patients with chronic hepatitis B (CHB). This prospective clinical and basic scientific study exclusively focuses on patients with the early antigen negative form of disease, which in developed countries is treated indefinitely with antiviral drugs. The investigators' study "BeNEG-DO," directly offers patients who are already taking standard oral Hepatitis B Virus (HBV) antiviral therapy for at least 192 weeks the option to stop or continue treatment. Drawing on data from pilot studies, including the investigators' own University of California, San Francisco and Sutter Institutional Review Board-approved study, the investigators will examine a finite HBV treatment strategy on clinical outcome and safety. In conjunction, the investigators will study immunologic mechanisms and gene expression profiles that correlate with and predict the post-treatment clinical course. The BeNEG-DO study could seriously question, and potentially change, the current treatment paradigm for millions of patients with CHB and also lead to new disease-terminating antiviral therapeutics.

DETAILED DESCRIPTION:
A prospective case-control study of safety and clinical outcomes, and of innate and adaptive immune responses and their genetic predictors, in adult human subjects with HBeAg-CHB who either continue or stop nucleoside or nucleotide analog (NA) antiviral therapy. Immune responses will be studied using liver tissue and serial peripheral blood samples. The immunological factors selected have been chosen based on preliminary and inferential evidence. Immunologic findings will be correlated with different serologic, virologic and biochemical outcomes. Genetic predictors of the type of response and respective clinical outcomes will also be sought.

ELIGIBILITY:
Inclusion Criteria:

1. HBeAg-CHB with at least 192 weeks (3.7 years) of complete viral suppression (serum HBV DNA <50 IU/ml) on NA therapy
2. No bridging fibrosis (≥ Metavir stage 3)
3. Normal liver tests and platelet count
4. Age 18-67
5. Otherwise healthy with no serious co-morbidities
6. Patients who are willing, prepared, and able to immediately resume antiviral treatment upon medical instruction and on satisfying study re-treatment criteria.

Exclusion Criteria:

1. HBeAg-CHB with virologic breakthrough while on NA therapy during the prior 192 weeks (3.7 years)
2. Age <18 or >67 years
3. Significant co-morbidities including co-infection and significant co-existing liver disease or anemia. Mild Non-Alcoholic Fatty Liver Disease (NAFLD) without Non-Alcoholic Steatohepatitis (NASH) or associated liver enzyme elevation will be allowed.
4. Bridging hepatic fibrosis (≥ Metavir stage 3) at the time of potential study entry

   a. Control Group: Determination will be based on historical biopsy data, imaging studies, Platelet count (<150,000), Aspartate aminotransferase to Platelet Ratio Index (APRI) <1.5) and Red Cell Distribution Width-to-Platelet Ratio (RPR) (<0.16) scores, and clinical assessment
5. Alanine Aminotransferase (ALT) above the quoted normal range
6. Clinical, serologic, radiological or biochemical suspicion for cirrhosis
7. Prior liver transplantation
8. A documented history of extrahepatic manifestations of hepatitis B, including renal disease and/or vasculitis
9. Cases: A family history of hepatocellular carcinoma due to hepatitis B virus in a first degree family member
10. On Prednisone or other immunosuppressive or immune-modulating therapy during the 6 months before study entry
11. Pregnancy
12. Patients who are not willing, prepared, and able to immediately resume antiviral treatment upon medical instruction and on satisfying re-treatment criteria

No one will be excluded on the basis of race, gender, religion, sexual orientation, or any cultural factor. An Institutional Review Board (IRB)-approved, translated consent will be used for patients that do not speak English

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2016-11-17 (Actual); Primary Completion 2026-05-25 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Serologic response and rate: HBsAg persistence versus loss; HBsAb production (+/-). This clinically relevant endpoint evaluates chronic HBV clearance and persistence | 10 years
  Annual seroclearance rates of 0.5%-0.8% in controls are assumed (American Association for the Study of Liver Diseases 2012 Poster 374) and equivalent to the estimated spontaneous rate (Hepatology 2009; 49:S45-55). In cases, 5-6% (based on Gastroenterology 2012 143:629:636) 5 year rates for HBsAg seroconversion (5%) or HBsAg loss only.

SECONDARY OUTCOMES:
Liver biochemical response: ALT level | 5 years
  These anticipated biochemical outcomes are based on Gastroenterology 2012 143:629-636
Virologic response: HBV DNA level | 10 years
  Hepatitis B Virus levels measured in International Units per milliliter
Case retreatment rate | 10 years
  As a measure of safety

CONTACTS AND LOCATIONS:
Overall Officials: Stewart L Cooper, MD, Principal Investigator — Sutter Health - California Pacific Medical Center; Jody L Baron, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - California Pacific Medical Center, San Francisco, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: Yes